CLINICAL TRIAL: NCT01478308
Title: Metformin With Standard Taxotere and Prednisone in the Treatment of Castration Resistant Prostate Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No accrual in initial period, PI decided to close study.
Sponsor: New Mexico Cancer Research Alliance (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INST 1011
Record Dates: First submitted 2011-09-02; First posted 2011-11-23 (Estimated); Last update posted 2013-03-06 (Estimated); Status verified 2013-03

CONDITIONS: Prostate Cancer
Keywords: prostate; castration resistant; hormone resistant; CRPC
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Metformin; Docetaxel; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Metformin hydrochloride — Metformin is administered orally, with food. Metformin tablets contain 500mg, 850mg, or 1000mg of metformin hydrochloride. Tablets contain inactive ingredients including pofidone and magnesium stearate. The coating for 500mg and 850mg tablets contains hypromellose. Metformin is an antihyperglycemic agent which decreases hepatic glucose production, decreases intestinal absorption of glucose, and improves insulin sensitivity by increasing peripheral glucose uptake and utilization.In this study, Metformin will be given 850 mg orally, with food, once daily for 1 week starting the week before first docetaxel infusion, and thereafter 850 mg twice daily.
Drug: Docetaxel — Docetaxel will be administered 75 mg/m2 as one hour infusion on day 1 every 21 days.
Drug: Prednisone — Prednisone will be given 5mg orally twice daily which is the standard regimen with docetaxel

SUMMARY:
This study is being conducted to determine the effectiveness of standard 3 weekly treatments using docetaxel and prednisone with metformin in patients with castration-resistant metastatic prostate cancer.

It is also being conducted to determine the levels of toxicity of metformin when added to every 3 weekly docetaxel treatments in patients with endocrine resistent, metastatic prostate cancer.

DETAILED DESCRIPTION:
This is a single-arm, non-randomized Phase II trial of docetaxel given every 3 weeks with metformin twice daily and Prednisone twice daily. The study duration of this trial is open ended. The patient would take the metformin only for as long as they are treated with docetaxel.

ELIGIBILITY:
Inclusion Criteria:

* All patients, 18 of age or older, with hormone refractory prostate cancer are eligible.
* Patients must have a life expectancy of at least 12 weeks.
* Patients must have a Zubrod performance status of 0-2.
* Patients must sign an informed consent.
* Patients should have adequate bone marrow function defined by an absolute peripheral granulocyte count of > 1,500 or cells/mm3 and platelet count >100,000/mm3 and absence of a regular red blood cell transfusion requirement.
* Patients should have adequate hepatic function with a total bilirubin < 2 mg/dl and SGOT or SGPT < two times the upper limit of normal, and adequate renal function as defined by a serum creatinine < 1.5 x upper limit of normal.
* Patients must have pathologically confirmed prostate cancer with PSA increasing despite androgen deprivation therapy.
* Diabetic patients on therapy with Metformin are eligible provided that their Metformin dose is at least 850mg twice daily.

Exclusion Criteria:

* Patients with symptomatic brain metastases are excluded from this study.
* Patients on insulin are not eligible.
* Patients may receive no other concurrent chemotherapy or radiation therapy during this trial.
* Patients with severe medical problems such as uncontrolled diabetes mellitus, cardiovascular disease, and congestive heart failure defined as New York Heart Association Class III or IV, hepatic dysfunction, or active infections are not eligible for this trial.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-06; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Measure efficacy | 7 years
  To determine the antitumor activity of metformin in combination with docetaxel and prednisone which are considered standard of care administered to patients with hormone refractory prostate cancer.

SECONDARY OUTCOMES:
Measure toxicity | 7 years
  To evaluate the quantitative and qualitative toxicities of metformin with this schedule, in this population

CONTACTS AND LOCATIONS:
Overall Officials: Richard Lauer, MD, Principal Investigator — University of New Mexico Cancer Center